CLINICAL TRIAL: NCT00218803
Title: A+ Asthma Rural Partnership
Brief Title: Teaching Children With Asthma and Who Live in a Rural Setting How to Self-Manage Their Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Arlene Butz, ScD, RN, MSN, Professor, Johns Hopkins University School of Medicine, Department of Pediatrics
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: HBV 99-01-11-01; 5R01NR005062-04 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Nurse asthma education intervention
- 2 (Other)
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Nurse asthma education intervention — Asthma Education
  Arms: 1
Behavioral: Control Group — Asthma Education
  Arms: 2

SUMMARY:
To determine if teaching rural children with asthma and their parents about appropriate medication use, asthma triggers unique to a rural setting and increasing access to medical care will result in a decrease in emergency department visits.

DETAILED DESCRIPTION:
Many self-management asthma interventions have demonstrated increase in asthma knowledge, reduced emergency department visits, increased self-efficacy and quality of life. The type of self-management interventions, specifically individualized and interactive educational interventions, have been suggested to have the strongest effect on asthma morbidity. Few studies have tested asthma self-management educational interventions in increasing knowledge, self-efficacy and quality of life in rural pediatric populations. The goal of this study was to test the effectiveness of an asthma educational intervention in improving asthma knowledge in rural children and their parent/caregivers. We hypothesized that an interactive asthma educational intervention would increase parent/caregiver and child asthma knowledge resulting in decreased emergency room visits in rural families of children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma, attend elementary school in rural county agreeing to participate

Exclusion Criteria: Participation in another asthma study or having other respiratory illness such as cystic fibrosis, BPD

-

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2000-08; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Decrease in emergency department visits | 10 months or 1 school year

SECONDARY OUTCOMES:
Asthma Education | 10 months or 1 school year

CONTACTS AND LOCATIONS:
Overall Officials: Arlene M Butz, SCD,MSN,BSN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Naumann PL, Huss K, Calabrese B, Smith T, Quartey R, Van de Castle B, Lewis C, Hill K, Walker J, Winkelstein M. A+ Asthma Rural Partnership coloring for health: an innovative rural asthma teaching strategy. Pediatr Nurs. 2004 Nov-Dec;30(6):490-4. PMID 15704600